CLINICAL TRIAL: NCT01176942
Title: Probiotics and Endotoxemia in Humans
Brief Title: Probiotics and Endotoxemia
Acronym: PROMS-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROMS-01
Record Dates: First submitted 2010-05-24; First posted 2010-08-06 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Metabolic Endotoxemia; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic bacterium Bifidobacterium lactis
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic bacterium Bifidobacterium lactis

INTERVENTIONS:
Dietary Supplement: Probiotic bacterium Bifidobacterium lactis — Probiotic placebo controlled intervention
  Other Names: Bifidobacterium animalis subsp. lactis

SUMMARY:
The purpose of this study is to determine whether probiotic treatment of overweight volunteers consuming high fat diet is able to reduce plasma lipopolysaccharide concentration.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 27 kg/m2; above 18 years of age
* Used to eat high fat diet (more than 40% of total energy intake)

Exclusion Criteria:

* Treated cardiovascular risk factors, treated hypertension, treated dyslipidemia, treated diabetes; Known diabetes, hypertension, dyslipidemia
* Severe illnesses
* Artificial heart valve
* Immunosuppression
* Regular consumption of probiotics
* History of bariatric surgery
* Consumption or wish to consume Orlistat
* Participation in other research
* Pregnancy or wishing/trying to get pregnant
* Inability to follow protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Level of plasma endotoxin (plasma levels of lipopolysaccharides) in the volunteers before and after the 12 week intervention | 12 weeks
  Quantitative, kinetic assay for the detection of gram negative bacterial endotoxin (lipopolysaccharide) is used to test whether the probiotic intervention can reduce plasma endotoxin levels (IU/ml) compared to the baseline.

SECONDARY OUTCOMES:
Volunteer weight before and after the 12 week intervention. | 12 weeks
Volunteer waist perimeter before and after the 12 week intervention | 12 weeks
Insulin resistance (HOMA-IR index), glycemia, insulinemia and glycated hemoglobin in the volunteers before and after the 12 week intervention | 12 weeks
  Insulin resistance (IR) will be quantified in the non-diabetic adults using the HOMA-IR index calculated as the product of fasting plasma insulin (in microunits per milliliter) and fasting plasma glucose (in millimoles per liter), divided by 22.5. Higher HOMA values indicate higher IR. Glycated haemoglobin is used as a biological measure indicator of blood glucose concentration over 3 months.
Brachial blood pressure of the volunteers before and after the 12 week intervention. | 12 weeks
Blood lipids in the volunteers before and after the 12 week intervention. | 12 weeks
  Plasma total cholesterol and triglycerides are measured by enzymatic methods. High-density lipoprotein (HDL) cholesterol is measured in the supernatant after sodium phosphotungstate/magnesium chloride precipitation. Low-density lipoprotein (LDL) cholesterol is determined by the Friedewald formula.
Serum inflammatory markers of volunteers before and after the 12 week intervention. | 12 weeks
  IL-6 (Interleukin-6) level is measured by an immunoenzymatic method, sCD14 is measured using an immuno-enzymatic method, and C reactive protein (CRP) levels is measured by an immunonephelemetric method.
Intestinal microbiota composition measured from stool samples before and after the 12 week intervention. | 12 weeks
  Stool samples are collected before and after the intervention and stored frozen until analysis. Bacterial DNA is extracted from the samples and relevant bacterial groups including genus Bifidobacterium, species Bifidobacterium animalis subsp. lactis, Enterobacteriaceae, Escherichia coli, Bacteroidetes and Lactobacillus are measures with quantitative real-time PCR.
Gut function questionaire as a measure of tolerability | Symptoms during last 6 days
  Questionaire is used to assess the tolerability of the probiotic supplementation. Questionaire includes questions on frequency and severity of flatulence and bloating, occurence of diarhea, frequency of defecation, and texture of feces using a stool chart.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Toulouse Hospital, Toulouse, Cedex 9, France